CLINICAL TRIAL: NCT01617174
Title: Observational Longitudinal Study of Pain in Men With Metastatic Castrate-Resistant Prostate Cancer
Status: Withdrawn | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Oregon Health and Science University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-110
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer
Keywords: prostate; pain assessment; 12-110
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- assessments completed by patients: A single-arm observational study will be conducted at three institutions in the Prostate Cancer Clinical Trials Consortium (PCCTC): Memorial Sloan-Kettering Cancer Center; Johns Hopkins; and Oregon Health & Science University. MSKCC is the coordinating center. The target enrollment is 400 patients, with at least 250 experiencing "moderate or worse" pain intensity at baseline, defined as a score of ≥4, the preferred regulatory cutoff.
  Interventions: Behavioral: Webcore telephone survey system

INTERVENTIONS:
Behavioral: Webcore telephone survey system — Patients will report pain and analgesic use through the automated telephone system, for 7 days in a row, once every 6 weeks. Data from diagnostic tests (CT Abdomen/Pelvis, Bone Scan, PSA, and circulating tumor cells) conducted during the study period will be collected from medical records by local personnel and entered into the secure online database quarterly, but no specific tests or schedules will be required in this observational study.

SUMMARY:
The first goal of this study is to learn more about the experience of pain and other symptoms in men being treated for advanced prostate cancer. The second goal of the study is to identify reliable ways of measuring pain which will be used in future clinical trials of treatments for advanced prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be ≥ 18 years old on the day of consent.
* The subject is able to understand written and spoken English.
* The patient must have histologically or cytologically confirmed prostate adenocarcinoma.
* The subject must have castration-resistant prostate cancer (CRPC).
* The subject must have metastatic disease involving bone, seen on radiographic imaging (bone scan, CT scan, PET scan, or MRI).
* The subject must be in a castrate state (e.g., currently receiving androgen deprivation therapy or have had an orchiectomy).
* The subject must be starting any line of systemic treatment post-androgen deprivation/antiandrogen therapy, with any of the following: chemotherapy (e.g., docetaxel, paclitaxel, carboplatin, cabazitaxel, or mitoxantrone); abiraterone acetate; MDV3100; ketoconazole; a clinical trial.
* The subject owns or has regular access to a telephone (cellular or land line).
* The subject is willing and able to self-report pain and analgesic use via an automated telephone system.
* The subject is willing and able to provide informed consent.

Exclusion Criteria:

* The subject has small cell or predominantly neuroendocrine differentiated prostate tumor.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be recruited from 3 different collaborating sites: MSKCC, John Hopkins, and OHSU. MSKCC will enroll approximately 200 patients, and John Hopkins and OHSU will each enroll approximately 100 patients; 400 participants will be enrolled in total. MSKCC is the coordinating site for this study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
pain score | 2 years
  Pain score changes will be correlated with each of the following: patient rating of change in pain, as well as changes in patient functional status, analgesic use, and various measures of disease status (imaging, PSA, circulating tumor cells). The distribution-based approach is to estimate meaningful change as one-half a standard deviation of the sample mean pain score.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/